CLINICAL TRIAL: NCT07051889
Title: TransfEr of the Lower Trapezius Tendon Versus Partial Cuff Repair Trial - TENET Trial
Brief Title: Lower Trapezius Tendon Transfer vs Partial Cuff Repair in Massive Rotator Cuff Tears
Acronym: TENET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Orthopaedic Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250033-01H
Record Dates: First submitted 2025-05-09; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Massive Rotator Cuff Tear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Trapezius Tendon Transfer (Active Comparator): The Lower Trapezius Tendon Transfer procedure involves transferring one of the other tendons located just outside the shoulder (the 'lower trapezius') and attaching this to the upper part of the arm bone, in the place of the torn rotator cuff tendon.
  Interventions: Procedure: Lower Trapezius Tendon Transfer
- Partial Rotator Cuff Repair (Active Comparator): The rotator cuff repair procedure involves reattaching the torn tendon(s) back to the upper part of the arm bone.
  Interventions: Procedure: Partial Rotator Cuff Repair

INTERVENTIONS:
Procedure: Lower Trapezius Tendon Transfer — This procedure is performed arthroscopically. The lower trapezius tendon is harvested from the back of the shoulder blade. A donor tendon is then used to extend the lower trapezius tendon so that it can reach the top of the arm bone. The tendon graft is then attached to the top of the arm bone, while the other end remains attached to the lower trapezius tendon itself. Any additional concomitant procedures (e.g. debridement, biceps release…etc.) may be performed as well.
  Arms: Lower Trapezius Tendon Transfer
Procedure: Partial Rotator Cuff Repair — This procedure is performed arthroscopically. The massive rotator cuff tear will be repaired by securing the loose tendon ends to the bone with suture anchors. The surgeon may also conduct a debridement of the area to remove any broken-down cartilage and tissues. Finally, the biceps tendon in will be further inspected for any damage or inflammatory changes, and the tendon may be released at the discretion of the surgeon (known as a biceps tenodesis or tenotomy depending on technique).
  Arms: Partial Rotator Cuff Repair

SUMMARY:
Very large tears of the shoulder tendons (the 'rotator cuff') that are not surgically repairable and in the absence of significant shoulder arthritis are common in older patients, and are associated with significant pain and functional limitations. Transfer of one particular tendon called the trapezius is becoming popular as a means of restoring function and improving pain in patients with massive rotator cuff tears. This tendon is appealing for transfer, as it has a similar line of pull to the infraspinatus (one of the rotator cuff tendons). There is currently no clear surgical consensus regarding the optimal treatment of patients with symptomatic massive irreparable rotator cuff tears that are appropriate candidates for joint salvage treatment, and no high level of evidence studies to guide clinical decision making have been published.

A pilot study is required prior to the development of a full-scale trial to assess its feasibility and recruitment across clinical sites, to determine protocol adherence (errors in randomization), and patient retention over a 12-month period.

The main objective of this pilot trial is to assess a composite measure of feasibility including recruitment, protocol adherence, and patient retention at one-year. The secondary objectives, currently exploratory only, are to determine the clinical outcomes of lower trapezius tendon transfer versus arthroscopic rotator cuff partial repair and biceps tenodesis/tenotomy on clinical outcome measures, shoulder function, adverse events and reoperation rates at two-years.

This pilot study is a parallel-group multicentre randomized controlled trial with participating sites across Canada, and one site in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and females over 18 years of age
* MRI confirmed diagnosis of massive rotator cuff tears defined using the Schumaier 2020 definition of massive cuff tears which includes the following criteria:

  * Retraction of the tendons to the glenoid rim, measured in either the coronal or axial plane
  * Greater than or equal to 67% of the greater tuberosity exposed in the axial plane
  * Diagnosed either with MRI or intra-operatively ** Note: patients may be screened for inclusion using ultrasound, and the Cofield or Gerber definitions of massive cuff tear defined as either 5cm or greater in maximum length or 2 more tendon involvement respectively, however their must meet the Schumaier et al 2020 definition for final inclusion.
* Features of irreparability of their rotator cuff tendon tear including:

  * Tendon retraction equal to or greater than 3cm16
  * Remnant tendon length of supraspinatus <15mm (as measured on coronal sequence of shoulder MRI)62
  * Goutallier grade 3 or 4 fatty infiltration of the supraspinatus
* An external rotation lag present on clinical exam. A positive external rotation lag will be considered as inability to perform external rotation with or against gravity.
* Provision of informed consent

Exclusion Criteria:

* Patients with complete subscapularis tears
* Patients with concomitant injuries of the affected shoulder
* Previous surgery on the affected shoulder
* Hamada grade 3 or above changes on plain films of the shoulder
* Substantial shoulder comorbidity (e.g. Bankart lesion or osteoarthritis [defined as joint space narrowing or osteophytes present on radiographs and confirmed at the time of arthroscopy])
* Substantial medical comorbidity that could impact the effectiveness of surgical intervention
* Inability to speak English or French
* Patients that will likely have difficulty with maintaining follow-up in the opinion of the evaluators (no fixed address, unwilling to be followed, incarcerated individuals, etc.)
* Cases involving litigation or workplace insurance claims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment and Follow-Up | 1-year
  Assess the feasibility of this pilot trial as determined by: (1) Recruitment rate of 6 per month across study centres; (2) 3 or fewer crossovers for enrolled participants; and (3) 85% of participants have a full adherence to protocol.

SECONDARY OUTCOMES:
The Western Ontario Rotator Cuff Score (WORC) | 2-years post-operative
  The WORC is a disease specific evaluation, proven to be an accurate and valid assessment of quality of life for rotator cuff disease. The WORC is a patient-reported measure, 21-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean a worse outcome.
Constant Score | 2-years post-operative
  The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points. The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES) | 2-years post-operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
Subjective Shoulder Value | 2-years post-operative
  A participant's subjective value on shoulder function will be assessed using a questionnaire. The overall functional value of the shoulder is written as a percentage from 0-100% of a normal shoulder. The higher the score, the better the outcome.
EuroQol EQ-5D-5L | 2-years post-operative
  The EQ-5D-5L quality of life questionnaire is a brief, easy to administer generic health status questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses (each question rated 1-5), lower scores indicate better outcome. It also includes a visual analogue scale for recording an individual's rating of their current health-related quality of life (scale 0 to 100), where a higher score indicates a better outcome.
Functional Range of Motion | 2-years post-operative
  Measured in degrees, and active movement. Range of motion measures include forward elevation (flexion), abduction, and external rotation from a neutral position, and internal rotation at the spinal level.
Strength | 2-years post-operative
  Measured using a dynamometer, and from the external rotation in neutral position. Strength will be reported in pounds.
Ultrasound | 1-year post-operative
  Ultrasound will be used to evaluate tendon healing rate after the repair or the transfer and assess for integrity. If the repair/transfer has healed it is considered a better outcome (tendon healing - yes/no).
Reoperation Rate | 2-years post-operative
  The number of reoperations will be monitored and recorded and compared between study groups. A higher rate of reoperations indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD FRCSC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be be shared with other researchers unless requested and an agreement is in place. Only aggregate data will be made public (overall study results).